CLINICAL TRIAL: NCT06606223
Title: A Study of Cases of Abnormal Serum Ammonia Attending Assiut University Children Hospital
Brief Title: A Study of Cases with Abnormal Serum Ammonia in Neonate and Children Attending Assiut University Children Hospital
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Menna Allah Sayed Mohamed sayed, Assistant Lecture, Assiut University
Other Study IDs: hyrerammoniamia
Record Dates: First submitted 2024-09-10; First posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Abnormal Serum Ammonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: serum ammonia test — precaution of withdrawal serum ammonia

SUMMARY:
To determine the etiology and clinical presentation of increased serum ammonia in infants and children presented to the Pediatric Genetic unit, Assiut University Hospital

-To study the effects of certain precautions on serum ammonia levels.

DETAILED DESCRIPTION:
Ammonia is an important source of nitrogen and is required for amino acid synthesis. Nitrogenous waste results from the breakdown and catabolism of dietary and bodily proteins, respectively. In healthy individuals, amino acids that are not needed for protein synthesis are metabolized in various chemical pathways, with the rest of the nitrogen waste being converted to urea. ammonium is excreted in the urine, resulting in net acid loss. The ammonia level generally remains low (<40 mmol/L) due to the fact that most ammonia produced in tissue is converted to glutamine. Glutamine is also excreted by the kidneys and utilized for energy production by gut cells, which convert the nitrogen byproduct into alanine, citrulline , and ammonia, which are transported to the liver via the bloodstream. Ammonia enters the urea cycle in hepatocytes or is ultimately converted to glutamine. Ammonia is toxic when present in high concentrations. Endogenous ammonia intoxication can occur when there is impaired capacity of the body to excrete nitrogenous waste, as seen with congenital enzymatic deficiencies. Patients with urea cycle defects (UCD), organic acidemias, fatty acid oxidation defects, bypass of the major site of detoxification (liver) (such as that seen in cirrhosis), can all present with elevations in ammonia. Ammonia diffuses through all body membranes, including the blood-brain barrier, and alters the amino acid pathway, ion transporters, and neuronal oxide reduction metabolism, with deleterious effect on neuron and astrocyte functioning.

Hyperammonaemia is defined as levels >110 µmol/L (198 µg/dL) in the neonatal period (including preterm) and >50 µmol/L (90 µg/dL) from that age onwards, The predominant clinical signs of acute hyperammonaemia are mostly due to cerebral oedema, They include irritability, rejection of feeds, vomiting or drowsiness in neonates and infants. In children, adolescents and adults, the main clinical signs are associated with differing degrees of acute encephalopathy: altered consciousness, ataxia, seizures, and coma Persistent or intermittent hyperammonaemia can produce chronic symptoms such as psychomotor delay or growth retardation. Older individuals can exhibit eating disorders or a wide spectrum of neuropsychiatric symptoms. In children, hyperammonaemia is often considered a metabolic derangement due to inborn errors of metabolism Such as organic acidemia, systemic carnitine deficiency, Reye syndrome, toxins, drug effect, or liver disease. On the other hand, if there is normal lactate and no metabolic acidosis associated with the hyperammonemia, then UCD, dibasic aminoaciduria, or transient hyperammonemia of the newborn are more likely. The association of elevated liver enzymes with hyperammonemia is most consistent after insult from hepatotoxins, Reye syndrome, or carnitine deficiency.

The severity of the clinical presentation depends on the peak ammonia level but is also influenced by the age of the patient, speed of onset or the presence of other underlying conditions. In many cases there is a triggering factor such as protein catabolism caused by prolonged fasting, fever, infections , gastrointestinal bleeding, dehydration, high protein intake, anesthesia, and surgery or use of specific medications. Ammonia level determination needs careful blood extraction and sample processing techniques because its levels easily rise when these requirements are not fulfilled (factitious hyperammonemia). The blood sample can be venous or arterial but needs to be drawn while the corresponding muscle group is at rest, without hypoxia (no compression or holding), and preferably through a large-caliber route to avoid hemolysis. The blood should be kept cold

ELIGIBILITY:
Inclusion Criteria:

* 1) Any neonate presented with Un explained

  1. Un controlled Convulsion
  2. Hypotonia
  3. Persistent neonatal Jaundice
  4. Persistent Metabolic acidosis
  5. Abnormal Urine Odour 2) Any Infant and Children Present With High Ammonia Level

Exclusion Criteria:

* Patient with (secondary) Non Metabolic Cause of Hyper ammonia

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Cohort descriptive studies
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
to determine the etiology and clinical presentation of increase serum ammonia in infant and children presented to the pediatric geneyic unit ,Assiut university Hospital | one year
  a. Inclusion criteria: Any neonate presented with Un explained
  1. Un controlled Convulsion
  2. Hypotonia
  3. Persistent neonatal Jaundice
  4. Persistent Metabolic acidosis
  5. Abnormal Urine Odour 2) Any Infant and Children Present With High Ammonia Level

IPD SHARING:
Plan to Share IPD: No